CLINICAL TRIAL: NCT00268580
Title: Evaluation of the Emergency Department Asthma Care Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Ontario Hospital Association (Other); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Dr. Diane Lougheed, Principal Investigator, Queen's University
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: DMED-782-04; ORS # 2003-342 (Other Grant/Funding Number: Government of Ontario)
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: Asthma; Care map; Clinical pathway; Education; Emergency department
MeSH Terms: conditions — Asthma; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Asthma care provided using care pathway
  Interventions: Behavioral: Asthma Care Pathway
- Control (No Intervention): Standard of care provided

INTERVENTIONS:
Behavioral: Asthma Care Pathway — Asthma care provided using standardized asthma care pathway
  Arms: Intervention

SUMMARY:
The purpose of the study is to evaluate whether the Emergency Department (ED) Asthma Care Project (ACP) leads to improved asthma care delivery and patient outcomes in the ED setting.

Hypothesis: Implementation of a multi-disciplinary asthma strategy/clinical pathway for the treatment of asthma in the ED, based upon the 1999 Canadian Asthma Consensus Guidelines (and subsequent updates), will increase adherence with published management guidelines in the ED setting, reduce variations in the emergency management of acute asthma, increase utilization of specialized asthma services and improve outcomes for patients following ED visits.

Methods:

This observational, pre- post-intervention study will compare a stratified sample of 10 Ontario hospital EDs (5 intervention and 5 control sites). Chart abstractions will be performed on all adult visits for acute asthma over a 3 month period before and after implementation of the Ontario Hospital Associations (OHA)'s (now Ontario Lung Association's (OLA's) ED Asthma Care Map. Patient and provider surveys and provider focus group post intervention will also be conducted. Primary outcome measures are hospitalizations and repeat ED visit rates. Secondary outcome measures include: length of stay in ED, self-reported adherence with referral to specialized asthma services made during index ED visit, self-reported asthma control, and use of self-management strategies (including use of action plan), use of asthma management strategies promoted by the care map (such as use of objective measure of airflow rates, use of steroids, education, referral to specialized asthma services on discharge). Ease of implementation and barriers to implementation will also be evaluated.

DETAILED DESCRIPTION:
Study findings may be used to support implementation of a standardized ED clinical pathway and related ED provider education program throughout Ontario.

Specific Objectives:

* To evaluate the impact of the pathway on patients.
* To evaluate the impact of the pathway on health care providers.
* To evaluate the ease of implementation of the pathway.

Study Design:

* Observational, pre- post-intervention study design.
* Comparison between intervention and control sites.
* Patient and provider surveys and provider focus group post intervention

Key Components:

1. Pre- and post- intervention chart abstraction of key elements of the process of asthma care in ED setting
2. Post-intervention telephone survey of patients
3. Post-intervention self-administered survey of health care providers
4. Post-intervention focus group

Methodology:

Background The Ontario Respiratory Outcomes Research Network (ORORN) is completing a Canadian Institutes of Health Research (CIHR)-funded study on "Determinants of Regional Variation in Emergency Department Utilization and Hospitalizations for Asthma in Ontario". This study included detailed chart abstractions on the process of care in the ED as well as detailed telephone questionnaires of adults and children who presented to EDs for treatment of acute asthma in a stratified sample of 14 hospitals across Ontario between March 2001 and Feb 2002. Data are available on over 5,000 ED visits. It is proposed that a number of these sites be approached to participate in ED ACP. A sub-set of data from these sites will provide baseline (pre-intervention) data, and some or all of the intervention and control sites for the ED ACP could be selected from the ORORN study sites. This would minimize (or potentially eliminate) costs of primary baseline data collection, and expedite collection of post-intervention data given the familiarity of sites and research personnel with the previous study instruments and protocol.

Selection of Intervention and Control Sites

Five intervention (Kingston General Hospital, Belleville General Hospital, Sudbury Regional Hospital, Renfrew Victoria Hospital, and Lake of the Woods District Hospital [Kenora]) and 5 control sites ( Prince Edward County Memorial Hospital, Lakeridge Hospital [Oshawa], St. Joseph's Hospital [Hamilton], Chatham District Hospital, and Owen Sound District Hospital) were selected. To ensure the sites are representative of Ontario, sites will be selected based upon a sampling frame which takes into consideration:

* Hospital/community size and location (urban/rural; geographic setting)
* Level of care (community/academic -tertiary/quaternary setting)
* Hospitalization rates for asthma in adults and children
* Presence of local specialized asthma services
* Access to quality baseline (pre-intervention) data from the ORORN ED study database
* Willingness of site to participate
* Location of other Asthma Plan of Action initiatives which might confound or be confounded by this intervention

Case identification within each ED will be performed by the method used by ORORN in a previous asthma ED study. This involves reviewing ED log books of presenting complaints potentially indicative of asthma OR electronically available data on disposition diagnoses of asthma. Potentially eligible patients will be approached as outlined below to obtain informed consent.

ED records (log books) from participating hospitals will be reviewed by a local research assistant for the preceding 24 to 72 hrs on a daily basis (Monday through Friday). Patient records with a chief complaint potentially indicative of an acute asthma exacerbation will be reviewed to capture all patients with a discharge diagnosis of an acute exacerbation of asthma. ED records with the following complaints in the logbook will be reviewed: asthma, shortness of breath, wheeze, cough, chest tightness, difficulty breathing. To be eligible the disposition diagnosis on the ED sheet must be asthma. Patients with a history of asthma presenting for reasons other than an acute exacerbation of asthma (such as prescription renewal or unrelated complaint) will be excluded.

Eligible patients will be mailed:

1. An introductory letter (Appendix A) outlining the purpose of the study, and informing them that they will be contacted by a research assistant within one week of their presentation to the hospital and invited to participate in the study and
2. A consent form (Appendix B). The Research assistant will contact patients by telephone to obtain informed consent. A telephone contact sheet (Appendix C) outlines the script to be used by the research assistant when speaking to potential participants. Once consent has been obtained the participant will answer a questionnaire (by telephone or in person). The questionnaire will be entered into a computerized version of a paper copy (Appendix D). The patient chart will then be abstracted also using a computerized version of the paper copy (Appendix E).

If the patient re-presents to the ED within 14 days of first visit the research assistant will contact the participant to obtain consent again. Any visit within the 14day period will be considered the same episode and repeat consent will not be required.

Pre-Intervention Chart Abstraction

Pre-intervention chart abstraction data will be obtained from either:

1. the ORORN ED study database, for sites that participated in the previous ORORN study, which contains data on adult and pediatric ED visits between March 2001 and February 2002, OR
2. retrospective primary data collection of ED visits for asthma between March 2001 and February 2002 for sites selected that did not participate in the previous ORORN ED study, utilizing the ORORN chart abstraction tool (or an abbreviated audit using specific components of that tool). (NOTE: If this is necessary, the research team and advisory committee will need to determine an appropriate abbreviated time-period to audit (eg. 3 months rather than a full 12 months) to remain within budget and meet target time-lines.)

Post-Intervention Chart Abstraction Post-intervention chart abstraction data will be obtained by primary data collection, using the ORORN chart abstraction tool (or an abbreviation thereof).

Post-Intervention Collection of Administrative Outcomes Hospitalization rates, readmission rates, and ED repeat visit rates for asthma and asthma-related conditions (as defined by the OHA Report Cards) will be obtained for each site directly or from national administrative databases (CIHI, NACRS). Referral rates to local specialized services will be collected where relevant and possible in small communities directly from the community resource involved.

Post-intervention Survey of Patients Patients eligible to participate will be mailed an introductory letter outlining the purpose of the study and a consent form. Subsequently, potential participants will be contacted by telephone by a research associate. After obtaining informed consent, a brief (5-10 minute maximum) telephone interview will be performed. A questionnaire for this purpose will be developed, including data elements from the ORORN regional variation study questionnaire to enable comparisons. It will also included whether the patient received education or referrals during their ED visit, whether they complied with referrals, and questions regarding the impact of the patient's visit on their asthma self-management skills and confidence.

Post-intervention Self-administered Survey of Health Care Providers A sample of ED health care providers involved in the delivery of aspects of the clinical pathway will be contacted at each site, and invited to complete a self-administered survey. A questionnaire for this purpose will be developed, to include perceived change in practice, perceived change in knowledge of recommended asthma management, perceived utility of the pathway, barriers to pathway implementation, and recommendations for improvement.

Post-intervention Site Representatives Focus Group

A post-intervention focus group including representatives from each participating site will be convened to gain additional insight into the site specific and aggregate outcomes and barriers that would be unlikely to emerge without the interaction found in a group. Aggregate data will be distributed to all sites, and site specific data to individual sites. The focus group will be invited to:

* assist with interpretation of quantitative findings;
* obtain perceptions of project outcomes and impacts;
* identify project strengths, weaknesses, and recommendations;
* identify solutions related to project implementation; and
* generate new ideas.

Ethical Considerations This study has been approved by the Queen's University Health Sciences and Affiliated Teaching Hospital's Research Ethics Board (REB) (Appendix F). Ethics is also being sought at all participating sites. The Queen's submission will be shared with sites and study coordinator will assist sites, where necessary, to facilitate the process.

Access to medical records will be sought from each institution. As this study involves questionnaire data collected by interview, stress may occur as a result of perceived pressure to answer specific questions. Participants will be informed during consent process that participation is voluntary, they may chose to not answer specific questions, and may withdraw from the study at any time without affecting their future medical care. Patient confidentiality will be ensured at all times. Confidential individual identification numbers will be randomly generated and sequentially by the web based data entry system, and used to link the abstracted data and questionnaire data.

Privacy officers have been contacted at each of the participating sites to ensure that the protocol meets the sites privacy protocol.

Potential Outcome Measures:

A. Impact of pathway on patients:

1. Hospitalization rate and length of stay
2. Length of stay in ED
3. Relapse rate to the ED for asthma, within 24 and 72 hours of ED visit
4. Self-reported adherence with referral to specialized asthma services made during index ED visit
5. Self-reported asthma control, and use of self-management strategies (including use of action plan)

B. Impact of the pathway on providers:

a. Use of Asthma Management Strategies Promoted by the ED ACP i. use of objective measure of airflow rates (PEFR or spirometry), and gas exchange (oxygen saturation, arterial blood gases) ii. types of asthma medications prescribed (bronchodilators, corticosteroids) in ED and upon discharge iii. route of medications prescribed (IV vs oral vs. inhaled steroids; metered-dose inhaler (MDI) vs nebulized bronchodilators) iv. documentation of assessment and teaching of device technique v. documentation of asthma action plan provision or revision vi. type of asthma education provided (e.g. environmental trigger avoidance, warning signs, medication use) vii. follow-up care recommendations or referrals (AEC, Asthma Clinic, Respirology Clinic, family physician) b. Utilization of Specialized Asthma Services i. referral rates (#/year) to local AECs and Asthma Clinics ii. types of providers involved in emergency asthma care

C. Ease of implementation of the pathway/ Barriers to implementation:

1. Proportion of patients enrolled on the ED ACP (Overall, by patient age category and by physician specialty)
2. Differences in patient demographics, physician demographics, day of week, time of day between patients enrolled vs. not enrolled
3. Perceived utility of pathway (overall, by site, and by profession)

ELIGIBILITY:
Inclusion Criteria:

* asthma plus or minus chronic obstructive pulmonary disease (COPD)
* ED visit for acute asthma treatment
* age 19 years or greater

Exclusion Criteria:

* COPD without asthma
* ED visit for asthma prescription renewal only

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-01; Primary Completion 2006-01 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
% of ED visitors admitted to hospital for asthma | At the end of the index ED visit (this is a dichotomous outcome. It is not possible to specify a "time frame").
  The patient is either admitted or not at the end of the ED visit.
Repeat Emergency Department visit rate for asthma | Within 24, 72h, 1 month

SECONDARY OUTCOMES:
Hospitalization length of stay | From ED presentation to hospital discharge
  It is not possible to specify a 'time frame'; the length of stay is the outcome
Length of stay in ED | From ED presentation to ED discharge
Self-reported adherence with referral to specialized asthma services made during index ED visit | At folllowup questionnaire
Self-reported asthma control, and use of self-management strategies (including use of action plan) | At followup questionnaire
Use of Asthma Management Strategies Promoted by the ED ACP: use of objective measure of airflow rates (PEFR or spirometry), and gas exchange (oxygen saturation, arterial blood gases) | During index ED visit (between ED presentation and ED discharge).
  These are dichotomous outcomes describing actual care received during the ED visit.
; types of asthma medications prescribed (bronchodilators, corticosteroids) in ED and upon discharge; route of medications prescribed (IV vs oral vs. inhaled steroids; MDI vs nebulized bronchodilators) | During index ED visit (between presentation and discharge, including discharge orders and instructions).
  These are dichotomous outcomes describing actual care received during the ED visit.
; documentation of assessment and teaching of device technique | During index ED visit (between ED presentation and ED discharge)
  During index ED visit (between presentation and discharge, including discharge orders and instructions).
; documentation of asthma action plan provision or revision | During index ED visit (between ED presentation and ED discharge)
; type of asthma education provided (e.g. environmental trigger avoidance, warning signs, medication use) | During index ED visit (between ED presentation and ED discharge)
; follow-up care recommendations or referrals (AEC, Asthma Clinic, Respirology Clinic, family physician) | During index ED visit (between ED presentation and ED discharge)
Utilization of Specialized Asthma Services | After discharge (within 12 months)
  Self-reported by patient on the followup questionnaire
; referral rates (#/year) to local AECs and Asthma Clinics | After discharge (within 12 months)
; types of providers involved in emergency asthma care | During index visit (between ED presentation and ED discharge)
Proportion of patients enrolled on the ED ACP (Overall, by patient age category and by physician specialty) | During index visit (between ED presentation and ED discharge)
Differences in patient demographics, physician demographics, day of week, time of day between patients enrolled vs. not enrolled | During index visit (between ED presentation and ED discharge)
Perceived utility of pathway (overall, by site, and by profession) | At time of followup survey (wihtin 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Diane Lougheed, MD, Principal Investigator — Queen's University
Locations (8):
- Canada (8):
  - Chatham Kent Health Alliance, Chatham, Ontario
  - Sudbury Regional Hospital, Greater Sudbury, Ontario
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Lake of the Woods District Hospital, Kenora, Ontario
  - Lakeridge Health Hospital, Oshawa, Ontario
  - Grey Bruce Health Services, Owen Sound, Ontario
  - Prince Edward County Hospital, Picton, Ontario
  - Renfrew Victoria Hospital, Renfrew, Ontario